CLINICAL TRIAL: NCT07235046
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel-group, Dose-finding Study to Evaluate Efficacy, Safety, and Tolerability of DII235 in Adults With Elevated Lipoprotein(a)
Brief Title: A Study of DII235 in Adults With Elevated Lipoprotein(a)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDII235A12201
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Lipoprotein Disorder
Keywords: Lipoprotein(a); cardiovascular disease; atherosclerotic cardiovascular disease (ASCVD); lipoprotein disorder; cardiovascular; cholesterol; hyperlipidemia; dyslipidemia; DII235
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis; Hyperlipidemias; Dyslipidemias | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: In order to preserve the integrity of the study and to minimize bias, a randomized double-blind study design is being used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm 1 (Placebo Comparator): Placebo
  Interventions: Drug: Saline
- Arm 2 (Experimental): DII235 dose 1
  Interventions: Drug: DII235
- Arm 3 (Experimental): DII235 dose 2
  Interventions: Drug: DII235
- Arm 4 (Experimental): DII235 dose 3
  Interventions: Drug: DII235
- Arm 5 (Experimental): DII235 dose 4
  Interventions: Drug: DII235

INTERVENTIONS:
Drug: DII235 — Solution for injection
  Arms: Arm 2; Arm 3; Arm 4; Arm 5
Drug: Saline — solution for injection
  Arms: Arm 1

SUMMARY:
The main purpose of this study is to determine the safety and efficacy of DII235 in adults with elevated lipoprotein(a).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study.
* Male or female participants 18 to 80 years of age (inclusive) at the screening.
* Lp(a) ≥ 150 nmol/L at screening, measured at the central laboratory.
* Participants with evidence of atherosclerotic cardiovascular disease and/or type 2 diabetes mellitus.

Exclusion Criteria:

* Severe renal dysfunction
* Hepatic dysfunction
* Malignancy within the last 5 years
* Use of investigational medications as defined in the protocol
* History or presence at screening of an underlying disease, or surgical, physical, medical, or psychiatric condition that, in the opinion of the Investigator, or sponsor if consulted, would potentially affect participant safety within the study or interfere with participating in or completing the study or with the interpretation of data

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2027-09-08 (Estimated); Study Completion 2028-09-08 (Estimated)

PRIMARY OUTCOMES:
Time averaged percentage change from baseline between Day 60 and Day 180 | baseline to day 60 and day 180
  Time averaged change from baseline in log Lp(a) measured between Day 60 and Day 180, defined as the area under the curve (AUC) between the Day 60 Visit date and the Day 180 Visit date, divided by the duration between the two visit dates.
Difference between DII235 dose 2 and placebo in time-averaged percent change from baseline in Lp(a) measured between Day 60 and Day 360 | baseline to day 60 and day 360
  Time averaged change from baseline in log Lp(a) measured between Day 60 and Day 360, defined as the area under the curve (AUC) between the Day 60 visit date and the Day 360 visit date, divided by the duration between the two visit dates.
Difference between DII235 dose 4 and placebo in time-averaged percent change from baseline in Lp(a) measured between Day 60 and Day 360 | baseline to day 60 and day 360
  Time averaged change from baseline in log Lp(a) measured between Day 60 and Day 360, defined as the area under the curve (AUC) between the Day 60 visit date and the Day 360 visit date, divided by the duration between the two visit dates.

SECONDARY OUTCOMES:
Difference between DII235 dose 1, dose 3 and placebo versus placebo in time-averaged percent change from baseline in Lp(a) measured between Day 60 and Day 360 | baseline to day 60 and 360
  Time averaged change from baseline in log Lp(a) measured between Day 60 and Day 360, defined as the area under the curve (AUC) between the Day 60 visit date and the Day 360 visit date, divided by the duration between the two visit dates.
Difference between DII235 doses versus placebo in time-averaged percent change from baseline in Lp(a) measured between Day 240 and Day 360 | baseline to day 240 and Day 360
  Time averaged change from baseline in log Lp(a) measured between Day 240 and Day 360, defined as the area under the curve (AUC) between the Day 240 Visit date and the Day 360 Visit date, divided by the duration between the two visit dates.
Difference between DII235 doses versus placebo with respect to the proportion of participants in achieving Lp(a) < 125 nmol/L at Day 180 and Day 360 | Day 180 and Day 360
  Participant's status of achieving Lp(a) < 125 nmol/L at Day 180 and at Day 360 (Yes, No), without having any defined intercurrent events.
Difference between DII235 doses versus placebo with respect to the proportion of participants in achieving Lp(a) < 75 nmol/L at Day 180 and Day 360 | Day 180 and Day 360
  Participant's status of achieving Lp(a) < 75 nmol/L at Day 180 and at Day 360 (Yes, No), without having any defined intercurrent events.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (43):
- United States (30):
  - Parkway Medical Center, Birmingham, Alabama
  - Heart Center Research Llc, Huntsville, Alabama
  - Cardiology and Medicine Clinic PA, Little Rock, Arkansas
  - National Heart Institute, Beverly Hills, California
  - Alliance Clinical, Canoga Park, California
  - Excel Medical Clinical Trials LLC, Boca Raton, Florida
  - Zenith Clinical Research, Hollywood, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Flourish Res Acq LLC North Miami, Miami, Florida
  - Inpatient Research Clinical LLC, Miami Lakes, Florida
  - Ocala Cardiovascular Research, Ocala, Florida
  - Cardiology Partners Clinical Research Institute, Wellington, Florida
  - Atlanta Heart Specialists LLC, Tucker, Georgia
  - AMR Chicago, Oak Brook, Illinois
  - Alliance for Multispecialty Research, Wichita, Kansas
  - CV Ins of the South, Lafayette, Louisiana
  - Metropolitan Cardiovascular Consultants Llc, Beltsville, Maryland
  - Anderson Medical Research, Ft. Washington, Maryland
  - Capitol Cardiology Associates, Lanham, Maryland
  - AA Medical Research Center, Flint, Michigan
  - AB Clinical Trials, Las Vegas, Nevada
  - K and R Research LLC, Marion, Ohio
  - TCV Clinical Studies, Linwood, Pennsylvania
  - Apex Cardiology Research Associates of Jackson, Jackson, Tennessee
  - Angiocardiac Care of Texas PA, Houston, Texas
  - Dallas Heart and Vascular Consultants PA, Houston, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - Northwest Houston Clinical Research PLLC, Tomball, Texas
  - Progressive Clinical Research, Bountiful, Utah
  - Dominion Medical Associates, Richmond, Virginia
- Germany (7):
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Potsdam, Brandenburg
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Gladbeck
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Münster
- Japan (6):
  - Novartis Investigative Site, Matsudo, Chiba
  - Novartis Investigative Site, Takamatsu, Kagawa-ken
  - Novartis Investigative Site, Miyhazaki, Miyazaki
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Shinjuku Ku, Tokyo
  - Novartis Investigative Site, Kyoto

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com